CLINICAL TRIAL: NCT03554044
Title: A Phase 1b Study of Talimogene Laherparepvec (T-VEC) in Combination With Chemotherapy or Endocrine Therapy in Patients With Metastatic, Unresectable, or Locoregionally Recurrent HER2-negative Breast Cancer
Brief Title: T-VEC With Chemotherapy or Endocrine Therapy in Treating Participants With HER2- Negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Jo Chien, Associate Clinical Professor, University of California, San Francisco
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17753; NCI-2018-00652 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2018-05-30; First posted 2018-06-12 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-03

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Estrogen Receptor Positive; HER2/Neu Negative; Invasive Breast Carcinoma; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8; Recurrent Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; exemestane; Fulvestrant; Letrozole; Paclitaxel; Taxes; talimogene laherparepvec; Tamoxifen; Albumin-Bound Paclitaxel; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort I (talimogene laherparepvec, chemotherapy) (Experimental): Patients receive talimogene laherparepvec intra-tumorally (IT) every 2 weeks for the first 10 weeks and every 3 weeks thereafter along with one of the following chemotherapies: paclitaxel (IV), nab-paclitaxel IV, or gemcitabine / carboplatin IV.
  Cycles repeat every 21 days until disease progression or unacceptable toxicity
  Interventions: Drug: Paclitaxel; Biological: Talimogene Laherparepvec; Drug: Nab paclitaxel; Drug: Gemcitabine; Drug: Carboplatin
- Cohort II (talimogene laherparepvec, endocrine therapy) (Experimental): Patients receive talimogene laherparepvec intra-tumorally (IT) every 2 weeks for the first 10 weeks and every 3 weeks thereafter along with letrozole PO, anastrazole PO, exemestane PO, tamoxifen PO on days 1-21 or fulvestrant IM every 2 weeks for 3 doses then every 4 weeks for the subsequent courses.
  Cycles repeat every 28 days until disease progression or unacceptable toxicity
  Interventions: Drug: Anastrozole; Drug: Exemestane; Drug: Fulvestrant; Drug: Letrozole; Biological: Talimogene Laherparepvec; Drug: Tamoxifen

INTERVENTIONS:
Drug: Anastrozole — Given PO
  Other Names: Arimidex; ICI-D1033; ZD-1033
  Arms: Cohort II (talimogene laherparepvec, endocrine therapy)
Drug: Exemestane — Given PO
  Other Names: Aromasin; FCE-24304
  Arms: Cohort II (talimogene laherparepvec, endocrine therapy)
Drug: Fulvestrant — Given IM
  Other Names: Faslodex; ICI 182,780; ZD9238
  Arms: Cohort II (talimogene laherparepvec, endocrine therapy)
Drug: Letrozole — Given PO
  Other Names: CGS 20267; Femara
  Arms: Cohort II (talimogene laherparepvec, endocrine therapy)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Cohort I (talimogene laherparepvec, chemotherapy)
Biological: Talimogene Laherparepvec — Given IT
  Other Names: ICP34.5-, ICP47-deleted Herpes Simplex Virus 1 (HSV-1) Incorporating the Human GM-CSF Gene; Imlygic; JS1 34.5-hGMCSF 47- pA-; T-VEC; OncoVEXGM-CSF
Drug: Tamoxifen — Given PO
  Other Names: Nolvadex
  Arms: Cohort II (talimogene laherparepvec, endocrine therapy)
Drug: Nab paclitaxel — Given IV
  Other Names: Abraxane
  Arms: Cohort I (talimogene laherparepvec, chemotherapy)
Drug: Gemcitabine — Given IV
  Other Names: Gemzar
  Arms: Cohort I (talimogene laherparepvec, chemotherapy)
Drug: Carboplatin — Given IV
  Other Names: Paraplatin
  Arms: Cohort I (talimogene laherparepvec, chemotherapy)

SUMMARY:
This phase Ib trials studies the side effects and how well talimogene laherparepvec works when given together with chemotherapy or endocrine therapy in treating patients with breast cancer that does not express the human epidermal growth factor receptor 2 (HER2) protein and has spread to other places in the body (metastatic), cannot be removed by surgery (unresectable), or has come back (recurrent). Biological therapies, such as talimogene laherparepvec, use substances made from living organisms that may attack specific tumor cells and stop them from growing or kill them. Chemotherapy drugs, such as nab-paclitaxel, gemcitabine, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Estrogen can cause the growth of breast cancer cells. Drugs used as endocrine therapy, such as letrozole, anastrozole, exemestane, tamoxifen or fulvestrant, may lessen the amount of estrogen made by the body or may may stop the growth of tumor cells by blocking estrogen from connecting to the cancer cells. Giving talimogene laherparepvec with chemotherapy or endocrine therapy may work better in treating patients with HER2-negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of intra-lesional talimogene laherparepvec injections in combination with chemotherapy or endocrine therapy in patients with metastatic, unresectable, or locoregionally recurrent HER2-negative breast cancer who have injectable sites of disease.

SECONDARY OBJECTIVES:

To evaluate the efficacy of talimogene laherparepvec in combination with chemotherapy or endocrine therapy in the study population

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT I (CHEMOTHERAPY): Patients receive talimogene laherparepvec intra-tumorally (IT) on day 1 of cycle 1, on days 1 and 15 of cycle 2, on day 8 of cycle 3, then on day 1 of subsequent cycles. Patients also receive paclitaxel or nab-paclitaxel intravenously (IV) over 60 minutes on days 1, 8, and possibly 15, or gemcitabine IV over 30-60 minutes and carboplatin IV over 30-60 minutes on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

COHORT II (ENDOCRINE THERAPY): Patients receive talimogene laherparepvec IT every 2 weeks for the first 10 weeks and then every 3 weeks thereafter. Patients also receive letrozole orally (PO), anastrazole PO, exemestane PO, tamoxifen PO on days 1-28 or fulvestrant intramuscularly (IM) every 2 weeks for 3 doses then every 4 weeks for the subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. Women or men 18 years or older with metastatic or locoregionally recurrent HER2-negative breast cancer. Resectable disease allowed.
2. Ability to understand and voluntarily sign informed consent prior to undergoing any study-related assessments or procedures, as well as adhere to the study visit schedule and other protocol requirements.
3. Histologic or cytologic confirmation of invasive breast cancer that is HER2-negative by standard clinical criteria.
4. Patients who will participate in the endocrine therapy cohort must have invasive breast cancer that is ER+ (>=1% ER staining by IHC).
5. At least one accessible and injectable lesion (ie. breast, chest wall, skin nodule or mass, axillary or supraclavicular lymph node) of at least 1cm. (Ultrasound imaging may be used as clinically indicated. Injection must be able to be performed at the bedside).
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
7. Concomitant use of bisphosphonates, RANKL antibody, and ovarian suppression is allowed.
8. Adequate organ function:

   * Absolute neutrophil count (ANC) >= 1.5x109/L for chemotherapy cohort, and >= 1.0x109/L for endocrine therapy cohort
   * Hemoglobin (Hgb) >= 9g/dL
   * Platelets (plt) >= 100 x 109/L for chemotherapy cohort, and >=75, 000 for endocrine therapy cohort
   * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <=2.5 x Upper Limit Normal (ULN). If liver metastases present <=5 x ULN allowed.
   * Serum total bilirubin <= 1.5 x ULN or direct bilirubin <= 1.5 × ULN in patients with well documented Gilbert's Syndrome
   * Serum creatinine <= 1.5 x ULN, or 24-hr clearance >= 60ml/min
   * International normalization ratio (INR) or prothrombin time (PT) or partial thromboplastin time (PTT)/ activated partial thromboplastin time (aPTT) <= 1.5 x ULN
9. Females of child-bearing potential (FCBP) should have a negative urine or serum pregnancy test within 72 hours prior to enrollment. If urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. FCBP must also be willing to adhere to acceptable forms of birth control (a physician-approved contraceptive method: tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) during the study treatment and through 3 months after the last dose of talimogene laherparepvec.

FCBP are defined as sexually mature women who:

* Have not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or,
* Have not been naturally postmenopausal for at least 12 consecutive months (i.e. has had menses at any time during the preceding 12 consecutive months)
* Must be willing to practice abstinence or use effective contraception for a minimum of 3 months following completion of study treatment (in addition to during study therapy).

Exclusion Criteria:

1. Any significant medical condition, laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
2. Any condition that confounds the ability to interpret data from the study.
3. Patients must have recovered from side effects resulting from prior cancer-directed therapy to a level of grade 1 or less (unless deemed not clinically significant by study investigator).
4. Symptomatic central nervous system metastases. Subjects with brain metastases that have been previously treated and are stable for 4 weeks after whole-brain radiotherapy (WBXRT) or 2 weeks after Stereotactic radiosurgery (SRS) are allowed. Patients must be stable off steroids for brain metastases for at least 7 days. Subjects with asymptomatic clinically insignificant brain metastases not requiring treatment are allowed. The exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
5. Patients with leptomeningeal disease.
6. History of symptomatic autoimmune disease or active autoimmune disease that has required systemic treatment in the 2 weeks prior to enrollment. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
7. Evidence of immune suppression due to: a) known human immunodeficiency virus (HIV) infection or AIDS; b) known leukemia or lymphoma; c) those who require high dose steroids (>10 mg/day of prednisone or equivalent within 7 days prior to enrollment) or other immunosuppressive therapies (>2weeks); d) active hepatitis B or C; e) congenital or acquired cellular and/or humoral immune deficiency; f) other signs or symptoms of immune system suppression or concurrent opportunistic infection.
8. Nab-paclitaxel arm: Grade 2 or higher neuropathy.
9. Known history of: cardiac disease, heart failure or decreased left ventricular ejection fraction, significant clinical arrhythmias.
10. Patients must not have received an investigational agent within 4 weeks or <= 5 half-lives, whichever is shorter, prior to starting study treatment.
11. Last dose of prior chemotherapy must be at least 2 weeks, and 2 weeks for targeted therapies, before first dose of study treatment. There is no required washout for endocrine therapy.
12. Major surgery or radiation ≤ 2 weeks prior to starting study treatment or who have not recovered from side effects of surgery or radiation.
13. Active herpetic skin lesions or prior complications of HSV-1 infection (e.g. herpetic encephalitis or keratitis).
14. Lesions with underlying infection or clinically meaningful bleeding.
15. Requires intermittent or chronic systemic (intravenous or oral) treatment with an antiherpetic drug (e.g. acyclovir), other than intermittent topical use. Patients requiring anti-herpetic prophylaxis during chemotherapy are excluded.
16. Previous treatment with talimogene laherparepvec or any other oncolytic virus.
17. Prior therapy with tumor vaccine.
18. Received live vaccine within 28 days prior to enrollment.
19. Known allergic reaction to talimogene laherparepvec, nab-paclitaxel, gemcitabine, carboplatin, aromatase inhibitors, tamoxifen, fulvestrant, or any of their components. An exception is made if the patient will not be receiving the offending agent/component (i.e. a patient who is allergic to nab-paclitaxel but will be receiving endocrine therapy is eligible).
20. Patients on therapeutic anticoagulation that cannot be held around injections.
21. Women who are pregnant or breast-feeding.
22. FCBP who are unwilling to use acceptable method(s) of effective contraception during study treatment and through 3 months after the last dose of talimogene laherparepvec.
23. Sexually active subjects and their partners unwilling to use a male or female latex condom to avoid potential viral transmission during sexual contact while on treatment and within 30 days after treatment with talimogene laherparepvec.
24. Subjects who are unwilling to minimize exposure with his/her blood or other body fluids to individuals who are at higher risks for HSV 1 induced complications (immunosuppressed individuals, HIV positive individuals, pregnant women, or children under the age of 1 year) during talimogene laherparepvec treatment and through 30 days after the last dose of talimogene laherparepvec.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment-related toxicities by maximum observed grade | Up to 2.5 years
  Treatment-related toxicities will be assessed according to NCI CTCAE v4.03, for all patients who receive at least one dose of study treatment. The distribution for the maximum observed grade for each adverse event will be tabulated and reported with 95% confidence interval
Maximum tolerated volume | Up to 2.5 years
  The maximum tolerated volume will be the highest volume (up to 4mL) that results in <=1 dose limiting toxicity (DLT) in 6 treated patients for the chemotherapy group. At least 15 patients will be treated in the chemotherapy cohort and at least 6 patients will be treated in the endocrine therapy cohort.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2.5 years
  The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence per Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1. Patients with complete response (CR) or partial response (PR) will be counted as having an objective response
Response duration | Up to 2.5 years
  Defined as the time from initial response to the first documented tumor progression.

CONTACTS AND LOCATIONS:
Overall Officials: Amy J Chien, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huppert LA, Gliwa AS, Tait M, Quintal L, Starzinski S, Cheung A, Moasser M, Majure M, Melisko M, Munster P, Rugo HS, Campbell M, Fong L, Chien AJ. Phase Ib study of intratumoral talimogene laherparepvec (T-VEC) in combination with chemotherapy or endocrine therapy in patients with advanced HER2-negative breast cancer. NPJ Breast Cancer. 2025 Nov 21;11(1):130. doi: 10.1038/s41523-025-00842-8. PMID 41271741